CLINICAL TRIAL: NCT04008095
Title: Evaluation of the Interest of PET/CT at 18F-FDG in the Post-therapeutic Management of Cervical Cancer at an Advanced Stage. Multicenter Prospective Observational Study
Brief Title: Interest of PET/CT at 18F-FDG in the Post-therapeutic Management of Cervical Cancer
Acronym: COLTEP
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: University Hospital, Brest (Other)
Responsible Party: Sponsor
Other Study IDs: 29BRC19.0084
Record Dates: First submitted 2019-05-31; First posted 2019-07-05 (Actual); Last update posted 2023-04-07 (Actual); Status verified 2023-04

CONDITIONS: Cervical Cancer
Keywords: cervical cancer; pet/ct; post-therapeutic; advanced stage; management
MeSH Terms: conditions — Uterine Cervical Neoplasms

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
A lot of studies have demonstrated the prognostic value of post therapy 18F-FDG PET/CT in the management of uterine cervical cancer. Post therapy 18F-FDG PET/CT is usually requested by a lot of clinicians.

Whereas 18F-FDG PET/CT is useful for prognosis in the follow-up, data are yet insufficient to clearly establish a formal recommendation.

This prospective multicenter observational study will evaluate the interest of post therapy 18F-FDG PET/CT in clinical management (within 2 months of treatment) in patients with cervical cancer at an advanced stage.

Main outcome :

The therapeutic impact of post therapy 18F-FDG PET/CT (within 2 months after the end of therapy) will be evaluated on the complete results included MRI.

Investigators will compare :

* decision of clinicians without 18F-FDG PET/CT results
* and decision of clinicians knowing entire results included results of 18F-FDG PET/CT.

DETAILED DESCRIPTION:
With approximately 3000 new cases estimated in France on 2017, the uterine cervical cancer is the twelfth cancer cause in women, responsible for 1000 deaths per year.

Management of uterine cervical cancer is well defined before treatment, especially for imaging including systematically pelvic MRI and 18F-FDG PET/CT.

A lot of studies have demonstrated the prognostic value of post therapy 18F-FDG PET/CT, due to semi quantitative parameters study, like the SUV max and delta SUV between pre and post therapy 18F-FDG PET/CT or qualitatively with the persistence of positive 18F-FDG PET/CT at the end of therapy.

Whereas 18F-FDG PET/CT is useful for prognosis in the follow-up, data are yet insufficient to clearly establish a formal recommendation.

Nevertheless, post therapy 18F-FDG PET/CT is still usually requested by a lot of clinicians.

Furthermore, the group of Parisian public hospital (AP-HP) has established a guide for the management of cervical cancer (2016) and recommends to systematically realize a 18F-FDG PET/CT after treatment for advanced cervical cancer.

Main purpose :

Evaluate the role of post therapy 18F-FDG PET/CT in clinical management (within 2 months of treatment) in patients with uterine cervical cancer at an advanced stage.

Main outcome :

The therapeutic impact of post therapy 18F-FDG PET/CT (within 2 months after the end of therapy) will be evaluated on the complete results included MRI.

Investigators will compare

* decision of clinicians without 18F-FDG PET/CT results
* and decision of clinicians knowing entire results included results of 18F-FDG PET/CT.

ELIGIBILITY:
Inclusion Criteria:

* Patient old ≥ 18 years
* Uterine cervical cancer with locally-advanced (FIGO 2019 IB3 to IVA)
* Histology: squamous cell carcinoma and adenocarcinoma
* Feasibility of a curative treatment
* Having formulated a non-opposition

Exclusion Criteria:

* Minor patient < 18 years
* Pregnancy or breastfeeding
* Other type of tumor than squamous cell carcinoma and adenocarcinoma
* FIGO 2019 < IB3 or > IVA
* Non-eligibility for the examination
* Contraindication to MRI and PET/CT
* Previous history of cancer
* Refusal of participation

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Gender Based: Yes
Study Population: Women recently diagnosed for an advanced cervical cancer (FIGO 2019 IB3 to IVA), and histologically proved.
Sampling Method: Probability Sample
Enrollment: 40 (Estimated)
Dates: Start 2020-01-08 (Actual); Primary Completion 2024-01-08 (Estimated); Study Completion 2026-01-08 (Estimated)

PRIMARY OUTCOMES:
The therapeutic impact of post therapy 18F-FDG PET/CT (within 2 months after the end of therapy) will be evaluated on the complete results included MRI. | Validated by six months follow up
  Investigators will compare
  * decision of clinicians without 18F-FDG PET/CT results
  * and decision of clinicians knowing entire results included results of 18F-FDG PET/CT.
  Gold Standard for the diagnosis of progression will be based on the conclusions of multi-disciplinary staff ruling on the results of composite data, including clinical examination, biology, histopathology, morphological imaging (MRI), functional imaging (PET/CT) and 6-month follow-up.
collection of the two décisions of RCP | Validated by six months follow up
  To make statistical analysis possible, the collection of the two decisions will be chosen from three cases of care envisaged below:
  1. Complete therapeutic response
  2. Equivocal response: doubt about the presence of residual disease.
  3. Strong suspicion of residual disease and/or progression Then, we will collect a percentage of patients with rightly changes on management induced by the result of the PET-CT at 18F-FDG.

SECONDARY OUTCOMES:
Physiological analysis parameter | 24 months follow up
  Diagnostic performances of PET/CT, Sensibility, Specificity, positive predictive value, negative predictive value
Prognostic factors | 24 months follow up
  Especially dynamic parameters (SUV max ...) and search for a statistical correlation between this value and PFS and OS.
Physiological analysis, hotspots study | 24 months follow up
  Hotspots study - Search for a density intersection between the local site residual disease of post-therapeutic 18F-FDG PET/CT and maximum-fixing tumor sites in 18F-FDG PET/CT Baseline.
Physiological analysis, hotspots study | 24 months follow up
  Hotspots study - Search maximum-fixing tumor sites in 18F-FDG PET/CT Baseline
Physiological analysis, hotspots study | 24 months follow up
  Assess the dosimetry of an escalation of the dose on these hotspots.

CONTACTS AND LOCATIONS:
Locations (2):
- France (2):
  - CHRU de Brest (Hôpital Morvan), Brest
  - Centre Henri Becquerel, Rouen

IPD SHARING:
Plan to Share IPD: Yes
All collected data that underlie results in a publication
Supporting Information: Study Protocol
Time Frame: Data will be available after the publication of result and ending three years maximum following the last visit of the last patient
Access Criteria: Data access requests will be reviewed by the internal committee of Brest UH. Requestors will be required to sign and complete a data accesss agreement